CLINICAL TRIAL: NCT03632356
Title: A Multi-Site Randomized Controlled Trial of a Stepped-Care Intervention for Emergency Department Patients With Panic Attacks and Panic Disorder
Brief Title: A Multi-Site RCT of a Stepped-Care Intervention for Emergency Department Patients With Panic Attacks and Panic Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Changi General Hospital (Other); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/2284
Record Dates: First submitted 2018-08-06; First posted 2018-08-15 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Panic Attacks and Disorders
MeSH Terms: conditions — Panic Disorder; Disease

STUDY DESIGN:
Intervention Model Description: 2 stage parallel group multi-site RCT design
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped Care Intervention (STEP) (Experimental): In a stepped-care model, all patients start with an evidence-based intervention of low intensity as a first treatment step. Progress is monitored and patients who do not respond adequately can subsequently be 'stepped up' to a higher intensity treatment. This model is now being recommended as the best strategy for treating panic attacks and panic disorder.
  Interventions: Behavioral: Stepped Care Intervention (STEP)
- Screening only (Active Comparator): Screening only for panic attacks and panic disorder using a gold standard clinical interview that provides coverage of the core symptoms of panic attacks and panic disorder.
  Interventions: Diagnostic Test: Screening only

INTERVENTIONS:
Behavioral: Stepped Care Intervention (STEP) — A stepwise progression of intervention according to the participant's response to the increasing levels of therapy. There will be 1 session of psychoeducation, followed by 5 sessions of Cognitive Behavioral Therapy (CBT) if panic symptoms do not improve at 1-month follow-up.
  Arms: Stepped Care Intervention (STEP)
Diagnostic Test: Screening only — Screening for probable panic attacks or panic disorder using the Structured Clinical Interview for DSM-5
  Arms: Screening only

SUMMARY:
Using a randomized controlled trial (RCT) design, the main objective of this study is to evaluate the clinical, patient-centered, and economic effectiveness of a stepped-care intervention for patients with panic attacks and panic disorder presenting to the busiest Accident and Emergency (A&E) departments of the largest public healthcare group in Singapore.

The RCT will have two arms: 1) treatment via an enhanced care pathway consisting of a stepped-care intervention for panic attacks and panic disorder; and 2) a control arm consisting of screening for panic attacks and panic disorder in the A&E and discharge (routine care). In addition to the baseline assessment, the study follow-up visits will occur at 1, 3, 6, and 12 months.

DETAILED DESCRIPTION:
Specific Aims and Hypotheses

Aim 1 (Primary): To evaluate the clinical effectiveness of a stepped-care intervention for A&E patients with panic attacks and panic disorder as compared to screening alone.

Aim 2: To evaluate the patient-centered effectiveness of a stepped-care intervention for A&E patients with panic attacks and panic disorder as compared to screening alone.

Aim 3: To evaluate the incremental cost-effectiveness of a stepped-care intervention for A&E patients with panic attacks and panic disorder compared to screening alone from the health system perspective.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 21+ years of age
3. Triage level 2 or 3
4. English or Mandarin speaking
5. Able to provide informed consent and read study materials
6. Presenting complaint of chest pain, palpitations, dizziness, or difficulty breathing
7. Score ≥ 3 on CDR screener
8. Diagnosis of panic attack or panic disorder confirmed on SCID interview
9. Willing to enter randomized trial

Exclusion Criteria:

1. Altered mental status (dementia, psychosis, substance intoxication/withdrawal)
2. Triage level 1
3. Non-English or Mandarin speaking
4. Unwilling or unable to complete study procedures
5. Symptoms of clear cardiac origin as determined by A&E physician
6. Deemed unfit due to possible adverse respiratory or cardiac outcomes by A&E physician
7. Clear organic cause for panic symptoms as evidenced by laboratory tests (FBC, UE, ECG, TROPONIN T, CXR)
8. Does not meet criteria for panic attack or panic disorder on SCID interview
9. Received CBT for panic symptoms in previous 12 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in panic scores at every 3 months from baseline using the Panic Disorder Severity Scale (PDSS; Shear et al., 2001) | Baseline, 1st month, 3rd month, 6th month, 12th month
  The PDSS is a 7-item semi-structured interview of panic symptom severity. Each item is rated on a 0 (none/mild) to 4 (extreme/severe) scale. A higher total score would represent severe panic symptoms.

SECONDARY OUTCOMES:
Short Form Health Survey (SF-36; Ware & Sherbourne, 1992) | Baseline, 1st month, 3rd month, 6th month, 12th month
  The SF-36 is a reliable and valid 36-item self-report questionnaire that evaluates multiple facets of health-related quality of life.
WHO Disability Assessment Schedule (WHO-DAS; World Health Organization, 2010) | Baseline, 1st month, 3rd month, 6th month, 12th month
  The WHO-DAS is a brief, cross-culturally valid, self-report questionnaire that is used to assess overall level of health and disability in clinical and general population settings.
Psychiatric Diagnostic Screening Questionnaire (PDSQ; Zimmerman & Mattia, 2001) | Baseline, 1st month, 3rd month, 6th month, 12th month
  The PDSQ is a reliable and valid self-report diagnostic questionnaire that has been widely used to assess the most common psychiatric disorders in outpatient settings.
EQ-5D (EuroQol Group, 1990) | Baseline, 1st month, 3rd month, 6th month, 12th month
  The EQ-5D is a patient self-report instrument that evaluates generic quality of life.

OTHER OUTCOMES:
Clinician Global Impression Severity Scale (CGI; Guy, 2008) | Baseline, 1st month, 3rd month, 6th month, 12th month
  The CGI is a clinician-rated instrument used to assess global severity of symptoms.The CGI ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). A higher total value indicates more severe panic symptoms and anxiety.
Panic Disorder Module of the Structured Clinical Interview for DSM-5 (SCID; First et al., 2015) | Baseline, 1st month, 3rd month, 6th month, 12th month
  The SCID is the gold standard tool for the reliable diagnosis of Axis I psychiatric disorders in clinical populations.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon C Sung, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shear MK, Rucci P, Williams J, Frank E, Grochocinski V, Vander Bilt J, Houck P, Wang T. Reliability and validity of the Panic Disorder Severity Scale: replication and extension. J Psychiatr Res. 2001 Sep-Oct;35(5):293-6. doi: 10.1016/s0022-3956(01)00028-0. PMID 11591432
- [Background] Guy, W., Clinical Global Impressions (CGI) Scale., In: Rush, A. J., First, M. B. and Blacker, D. (eds), Handbook of Psychiatric Measures, Washington, D.C.: American Psychiatric Publishing, Inc., 2008.
- [Background] First, M. B., Williams, J. B. W., Karg, R. S. and Spitzer, R. L., Structured Clinical Interview for DSM-5 Disorders-Clinician Version (SCID-5-CV), Arlington, VA: American Psychiatric Association, 2015.
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] World Health Organization, Measuring Health and Disability: Manual for WHO Disability Assessment Schedule - WHODAS 2.0, Geneva, 2010.
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Sung SC, Rush AJ, Earnest A, Lim LEC, Pek MPP, Choi JMF, Ng MPK, Ong MEH. A Brief Interview to Detect Panic Attacks and Panic Disorder in Emergency Department Patients with Cardiopulmonary Complaints. J Psychiatr Pract. 2018 Jan;24(1):32-44. doi: 10.1097/PRA.0000000000000283. PMID 29320381
- [Background] Zimmerman M, Mattia JI. A self-report scale to help make psychiatric diagnoses: the Psychiatric Diagnostic Screening Questionnaire. Arch Gen Psychiatry. 2001 Aug;58(8):787-94. doi: 10.1001/archpsyc.58.8.787. PMID 11483146
- [Derived] Sung SC, Lim L, Lim SH, Finkelstein EA, Chin SLH, Annathurai A, Chakraborty B, Strauman TJ, Pollack MH, Ong MEH. Protocol for a multi-site randomized controlled trial of a stepped-care intervention for emergency department patients with panic-related anxiety. BMC Psychiatry. 2022 Dec 16;22(1):795. doi: 10.1186/s12888-022-04387-z. PMID 36527018